CLINICAL TRIAL: NCT03963869
Title: A Quasi-Experimental Study to Assess the Effectiveness of Malaria Camps as Part of the Odisha State Malaria Elimination Drive
Brief Title: Effectiveness of Malaria Camps as Part of the Odisha State Malaria Elimination Drive
Acronym: CSCMi20
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Community Welfare Society Hospital (Unknown); Martin Luther Christian University (Unknown); Indian Institute of Public Health, India (Other); National Institute of Research in Tribal Health (Unknown); National Vector Borne Disease Control Programme (Unknown); University Hospital, Umeå (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); New York University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 19-00122
Record Dates: First submitted 2019-05-22; First posted 2019-05-28 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Intervention Model Description: Quasi-experimental cluster-assigned stepped-wedge study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A: New Malaria Camp (MC) village (Experimental): Receives MC intervention in year 1 and year 2.
  Each individual will be followed up 3 times (baseline and follow-ups 1, 2, and 3; 4 visits per individual) in the 2 year time frame of phase 1.
  Interventions: Other: Malaria Camps
- Arm B: No Malaria Camp (MC) village (Active Comparator): Receives Standard Malaria Control in Year 1 and MC intervention in Year 2.
  Each individual will be followed up 3 times (baseline and follow-ups 1, 2, and 3; 4 visits per individual) in the 2 year time frame of phase 1.
  Interventions: Other: Malaria Camps
- Arm C: Old Malaria Camp (MC) village (Active Comparator): Villages already in receipt of MCs prior to study initiation to study longer term effects.
  Each individual will be followed up 3 times (baseline and follow-ups 1, 2, and 3; 4 visits per individual)) in the 2 year time frame of phase 1.
  Interventions: Other: Malaria Camps

INTERVENTIONS:
Other: Malaria Camps — The Govt. of India Malaria Control Programme (MCP) of Odisha provides ITNs and IRS, and trains community health workers (ASHAs) on the diagnosis and treatment of malaria, providing them with antimalarial drugs so that malaria treatment is available even in remote villages. Faced with a persistent burden of malaria in forest villages, the MCP recently introduced malaria camps (MCs) combining focused screening and treatment in villages with intensified vector control. The program includes one round of testing and treatment for the whole village population before the monsoon season, followed by one round of screening and treating of fever cases only during the monsoon season.

SUMMARY:
The Odisha State Malaria Control Program (India) has introduced 'malaria camps' where teams of health workers visit villages to educate the population, enhance vector control with long-lasting insecticide nets (LLINs) and indoor residual spraying (IRS), and perform village-wide screening with rapid diagnostic tests and treatment for malaria. The long-term goal of this project is to evaluate the effectiveness of malaria camps (MCs) by determining if they reduce malaria, and to characterize malaria transmission in MCs.

DETAILED DESCRIPTION:
The persistently high malaria burden in the remote forested areas of Odisha, India has led to the introduction of 'malaria camps' by the Odisha State Malaria Control Program where teams of health workers visit villages to educate the population, enhance vector control with long-lasting insecticide nets (LLINs) and indoor residual spraying (IRS), and perform village-wide screening with rapid diagnostic tests and treatment for malaria. The camps appear to be very effective but this is hard to assess in the context of ongoing changes such as LLIN introduction. The long-term goal of this project is to evaluate the effectiveness of malaria camps (MCs) by determining if they reduce malaria, and to characterize malaria transmission in MCs. The major objective to achieve this is through a quasi-experimental study (i.e., pretest-post-test control group design) of the effectiveness of the intervention, to determine if MCs reduce the prevalence of clinical and asymptomatic malaria as detected by PCR. In the first year, villages will be assigned across three study arms: arm 1 to receive new MCs; arm 2 is a control with no MCs but with standard malaria control; and arm 3 consists of villages already in receipt of MCs to study longer term effects. In the second year, both arm 1 and arm 2 villages will receive the intervention (i.e., a non-randomized stepped-wedge design). MC effectiveness will be evaluated from epidemiologic surveys and PCR detection of malaria prevalence with and without MCs.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent by individuals greater than 17 years old, or consent by a parent/guardian of children 1-6 years old, or assent of individuals from 7-17 years old along with consent from his or her parent or legal guardian.
* A complete understanding of study procedures/protocols, as delineated in the consent and assent forms and information sheets.
* Individuals have the ability and are willing to comply with study procedures for the entire length of the study.

Exclusion Criteria:

* Individuals less than 12 months or more than 69 years of age will be excluded.
* Persons who do not understand the study or are physically unable to make monthly visits.

Ages: 1 Year to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2463 (Actual)
Dates: Start 2019-08-03 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Parasite presence | 24 Months
  The standard molecular method of (conventional) PCR + gel electrophoresis will be used to measure parasite presence. All reactions are run with Plasmodium positive controls and negative controls. 10% of samples are QC-ed at second independent site.
  The results can be continuous and categorical. Continuous variables will be transformed into categorical variables, so that infections can be sub-divided into symptomatic or asymptomatic.
Parasite species | 24 months
  The standard molecular method of (conventional) PCR + gel electrophoresis will be used to measure parasite species. All reactions are run with Plasmodium positive controls and negative controls. 10% of samples are QC-ed at second independent site.

SECONDARY OUTCOMES:
Malaria as detected by RDT | 24 months
  Malaria as detected by a rapid diagnostic test
Gametocyte density | 24 Months
  Measured by quantifying the number of gametocyte infected erythrocytes and dividing by the number of leukocytes or by quantitative reverse transcriptase real time PCR. Both results can be measured continuously and categorically (data will be transformed). To account for a mixed-infection (either by species or by multiple strains) we will take the gametocyte to trophozoite ratio to reduce any apparent bias.
Hemoglobin | 24 months
  Hemoglobin will be measured by POC testing which provides both continuous and categorical data (when analyzed by local standards) regarding anemia status.
BMI | 24 months
  Height in cm will be measured with a height measuring tape. Weight in kg will be measured with a scale. Participants will be asked to remove shoes and shawls or cardigans, or other clothing that can be removed without ethical concerns.
  BMI will be calculated as (kilograms/meters squared). Measures will be adjusted by age using the WHO Multicentre Growth Reference Study Group's 2006 WHO Child Growth Standards: Length/height-for-age, weight-for-age, weight-for-length, weight-for-height and body mass index-for-age: Methods and development.
  Categorical BMI measurements will be based on standards for Asian Indians: Misra A, Chowbey P, Makkar BM, et al. Consensus Statement for Diagnosis of Obesity, Abdominal Obesity and the Metabolic Syndrome for Asian Indians and Recommendations for Physical Activity, Medical and Surgical Management.
Body temperature | 24 months
  Body temperature will be measured with a digital thermometer placed under the participant's tongue reported in degrees Fahrenheit.
Mid-upper arm circumference | 24 months
  Mid-Upper Arm Circumference (MUAC) Mid-Upper Arm Circumference (MUAC) is the circumference of the left upper arm, measured at the mid-point between the tip of the shoulder and the tip of the elbow (olecranon process and the acromium). Participants will be asked to remove any clothes that may hinder the measurement (preferable directly on skin, but tight clothes can be accepted if they are difficult to remove).
  MUAC will be measured in cm to one decimal using a Myotape/tape measure.
Plasmodium-specific serology | 24 months
  Measured by a high-throughput bead-based cytometric assay provides continuous and categorical (seropositive vs. seronegative) results.
Plasmodium parasite genomic epidemiology | 24 months
  Plasmodium infections will be characterized for their mixed clonality, genetic diversity, and molecular force of infection by MinIon or Illumina NextGen sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Jane Carlton, PhD, Principal Investigator — New York University
Locations (1):
- Community Welfare Society Hospital, Rourkela, Odisha, India

IPD SHARING:
Plan to Share IPD: Undecided
Historically we submit all of our data to public databases.

DOCUMENTS (1):
  • Informed Consent Form (2019-03-01): https://cdn.clinicaltrials.gov/large-docs/69/NCT03963869/ICF_000.pdf